CLINICAL TRIAL: NCT00780390
Title: Autonomic Dysfunction and Spinal Cord Stimulator in Complex Regional Pain Syndrome
Brief Title: Autonomic Dysfunction and Spinal Cord Stimulation in Complex Regional Pain Syndrome
Acronym: CRPS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment and discontinued funding
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 071060; CTSA 1 UL 1 RR024975 NCRR/NIH
Record Dates: First submitted 2008-05-08; First posted 2008-10-27 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Complex Regional Pain Syndrome
Keywords: RSD; SCS; CRPS; Complex regional pain syndrome patients before undergoing spinal cord stimulator implant and under other treatments
MeSH Terms: conditions — Complex Regional Pain Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRPS patients without spinal cord stimulation (Placebo Comparator): CRPS patients declining spinal cord stimulation therapy. Autonomic Function will be assessed at baseline and again within 2 years.
  Interventions: Other: Autonomic Function Assessment
- CRPS patients: candidates for spinal cord stimulator (Experimental): CRPS patients who are candidates for spinal cord stimulator implant. These patients will have Autonomic Function assessments before and after the Standard of Care spinal cord stimulation implant
  Interventions: Other: Autonomic Function Assessment

INTERVENTIONS:
Other: Autonomic Function Assessment

SUMMARY:
To demonstrate that spinal cord stimulator has an effect on sympathetic function (the one that give us the fight and flight response). Therefore, if the spinal cord stimulator has an effect on sympathetic function, the responses from CRPS patients to different stimuli will differ significantly pre and post SCS implant.

If CRPS patients exhibit autonomic, CRPS patients could be stratified according to their sympathetic function pre-implant. It is expected that patients with a moderate/mild form of autonomic dysfunction will have better outcomes with the SCS.

DETAILED DESCRIPTION:
Currently the mechanisms of Complex Regional Pain Syndrome (CRPS) are poorly understood and stratification of either diagnosis or therapy is very weak. . There is a great need to develop and validate more objective methods to characterize and stratify CRPS that better diagnostic and therapeutic approaches are available. Spinal Cord Stimulation (SCS) has been used as the last resource to alleviate pain and re-establish function in CRPS patients. However, there is a disagreement over how it works. An underlying concept is that it works by modulating autonomic nervous system (ANS) activity. Therefore, ANS parameters could be useful to stratify patients. Our preliminary studies indicated that SCS has also an effect on blood pressure regulation and improves the CRPS patients' response to Valsalva maneuver -a test of autonomic function. The Autonomic Nervous System function in adult CRPS patients has not yet been studied. The only existing study of CRPS and autonomic function showed that 15% of the patients suffer from syncope and increased heart rate during upright position similar to same aged patients with postural tachycardia syndrome - a syndrome of autonomic dysfunction. It is unclear if autonomic dysfunction is present in CRPS patients because ANS activity is altered by chronic pain or whether or not ANS activity contributes to CRPS. Therefore, we proposed to study the autonomic function in CRPS patients by standardized autonomic function and to evaluate the effect of the SCS on autonomic function in CRPS patients before and after spinal cord stimulator implant. This is a 24 months study.

ELIGIBILITY:
Inclusion Criteria:

* CRPS patients meeting the inclusion criteria according to the International Association for the Study of pain task Force will be included in the study.
* Age: 18 to 65.
* Disease duration of at least 6 months.
* History of unsuccessful long lasting therapies: physical therapy, transcutaneous electrical stimulation and medication.

Exclusion Criteria:

* Presence of current or past pulmonary, hepatic, renal disease, arthritis, hematopoietic, and neurological diseases not related to CRPS.
* Anticoagulant therapy, cardiac pacemaker used.
* Pregnancy test for females is positive.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Change in muscle sympathetic nerve activity | At baseline and within 2 years

SECONDARY OUTCOMES:
Heart rate and blood pressure responses | At baseline and within 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Konrad, M.D., Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States